CLINICAL TRIAL: NCT07118228
Title: Evaluation of the Relationship Between Ultrasonographic Muscle Morphology, Functional Properties, and Clinical Parameters in Children With Spastic Cerebral Palsy
Brief Title: Ultrasonographic Assessment of Muscle Morphology, Function, and Clinical Findings in Spastic Cerebral Palsy
Acronym: US-sCP
Status: Recruiting | Type: Observational
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Nigar Dursun, Principal Investigator, Department of Physical Medicine and Rehabilitation, Kocaeli University
Other Study IDs: 2025/301; GOKAEK-2025/15/08 (Other: Kocaeli University Non-Interventional Clinical Research Ethics Committee)
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Muscle Spasticity; Gait Disorders, Neurologic; Cerebral Palsy, Spastic
Keywords: Spastic Cerebral Palsy; Muscle Morphology; Shear Wave Elastography; Muscle Architecture; Superb Microvascular Imaging; Muscle Stiffness; Pennation Angle; Fascicle Length; Intramuscular Vascularity; Echo Intensity; GMFM-66; Gross Motor Function; Muscle Morphology and Function; Ultrasound Imaging; Ultrasound Imaging of Spastic Muscle; Functional Assessment
MeSH Terms: conditions — Muscle Spasticity; Gait Disorders, Neurologic; Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Spastic CP Cohort: Ambulatory children with spastic cerebral palsy classified within GMFCS levels I to III. Participants undergo clinical and ultrasound-based assessments to evaluate muscle morphology, functional properties, and their relationship with motor function.

SUMMARY:
This study focuses on children with spastic cerebral palsy and aims to examine how muscle morphology and tissue characteristics, as assessed by ultrasound, may relate to functional motor abilities. It is designed as a prospective, cross-sectional, observational study. Planned ultrasound-based assessments include parameters such as muscle thickness, pennation angle, fascicle length, echo intensity, tissue stiffness (via shear wave elastography), and microvascular flow (via superb microvascular imaging). These measurements are intended to be compared with standard clinical evaluations, including the GMFCS, GMFM-66, MAS, MACS, and Tardieu Scale. The study seeks to contribute to a better understanding of the relationship between muscle architecture and functional outcomes, with the goal of generating insights that may inform individualized rehabilitation planning.

DETAILED DESCRIPTION:
This prospective, cross-sectional observational study aims to explore the relationship between ultrasonographically assessed muscle morphology, functional muscle characteristics, and standardized clinical parameters in ambulatory children diagnosed with spastic cerebral palsy (CP). The research seeks to enhance the understanding of muscle structure-function relationships in this population, with the broader goal of contributing to personalized rehabilitation strategies and clinical decision-making.

Cerebral palsy is a non-progressive neurodevelopmental disorder resulting from brain injury or maldevelopment during the prenatal, perinatal, or early postnatal period. Spastic cerebral palsy is the most common subtype, characterized by upper motor neuron lesions that lead to increased muscle tone, spasticity, and movement dysfunction. These neuromuscular alterations often result in secondary changes in muscle morphology, such as increased stiffness, reduced muscle volume, shortened fascicle length, altered fiber orientation, and impaired microcirculation. Understanding how these changes relate to functional limitations remains an important goal in pediatric rehabilitation research.

In this study, both structural and functional properties of skeletal muscles are planned to be assessed using a combination of high-resolution ultrasound techniques. The targeted muscles for assessment include one lower limb and one upper limb muscle: the medial gastrocnemius and the brachialis. These muscles were selected due to their relevance in gross motor and upper limb function in children with spastic CP.

The ultrasonographic parameters planned for evaluation include muscle thickness (MT), fascicle length (FL), pennation angle (PA), cross-sectional area (CSA), and echo intensity (EI). Additionally, muscle stiffness will be estimated through shear wave elastography (SWE), and vascularity will be evaluated using superb microvascular imaging (SMI) or a similar non-contrast-enhanced microvascular ultrasound technique. These advanced imaging modalities allow for the assessment of tissue elasticity and intramuscular blood flow, serving as potential surrogate markers of muscle quality and pathology.

Measurements will be acquired under standardized conditions, with the muscles in a relaxed state and proper anatomical alignment. Multiple images and repeated measurements will be obtained to ensure consistency. Longitudinal and transverse imaging planes will be used depending on the parameter being evaluated. The ultrasonographic protocol is designed to minimize operator-dependent variability and to ensure reproducibility across participants.

Clinical assessments will be conducted using standardized functional and spasticity-related scales. Gross motor function will be evaluated using the Gross Motor Function Classification System (GMFCS) and the Gross Motor Function Measure-66 (GMFM-66). Hand function will be categorized using the Manual Ability Classification System (MACS). Spasticity will be evaluated through the Modified Ashworth Scale (MAS) and the Tardieu Scale, which include assessments of the angle of muscle reaction (R1), passive range of motion (R2), and their difference (R2-R1). Where applicable, additional tools such as the Assisting Hand Assessment (AHA) and the Observational Gait Scale (OGS) may be employed to further characterize upper limb use and gait function.

Eligible participants include children aged 4 to 18 years with a diagnosis of spastic cerebral palsy, classified within GMFCS levels I to III. Children with recent exposure to interventions that could alter muscle morphology, such as botulinum toxin injection (within 6 months) or orthopedic surgery, will be excluded. Other exclusion criteria include the presence of non-spastic CP subtypes, neuromuscular disorders unrelated to CP, or inability to cooperate with assessments. All assessments will be performed in a single visit, without any therapeutic intervention being administered as part of the study.

The study involves no invasive procedures and is considered minimal risk. Its aim is descriptive and correlational, without testing any treatment or hypothesis regarding clinical efficacy. A power analysis was conducted to determine the required sample size for detecting statistically significant correlations. Ethical approval has been obtained from the relevant institutional ethics board. Data collected from participants will be anonymized and managed according to institutional and national data protection guidelines.

Planned statistical analyses include correlation coefficients between imaging parameters and clinical scores, along with regression analyses to identify potential predictors of motor function. Subgroup analyses may explore differences based on GMFCS level, age, or previous therapy exposure. The findings may provide insights into the associations between muscle architecture and clinical function in children with spastic CP, contributing to the development of individualized rehabilitation protocols and improved clinical monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of spastic cerebral palsy (SCP) according to the criteria defined by Rosenbaum et al. (2007)
* Age between 4 and 18 years
* Gross Motor Function Classification System (GMFCS) Level I, II, or III
* Manual Ability Classification System (MACS) Level I, II, III, or IV

Exclusion Criteria:

* Non-spastic types of cerebral palsy (e.g., dyskinetic, ataxic)
* Diagnosis of neuromuscular disorders other than cerebral palsy (e.g., hereditary neuropathy, myopathy)
* Presence of muscle contractures or fixed deformities in the limbs selected for ultrasound and clinical assessment
* Cognitive or behavioral impairments that prevent cooperation during ultrasound or clinical evaluation
* Botulinum toxin-A (BoNT-A) injection applied to the target muscles within the last 6 months
* Current treatment with oral or intrathecal antispastic medications
* History of orthopedic surgery or selective dorsal rhizotomy involving the target muscles
* Acute infection, febrile illness, or severe systemic disease (e.g., advanced heart failure, respiratory insufficiency) that may compromise the safety of assessments

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Ambulatory children aged 4 to 18 years diagnosed with spastic cerebral palsy, classified within GMFCS levels I-III and MACS levels I-IV, who are referred to a pediatric rehabilitation clinic for routine evaluation and are eligible for non-invasive ultrasound-based muscle morphology and clinical assessments.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Relationship between muscle morphology parameters and motor function in children with spastic cerebral palsy | At baseline (single assessment session)
  This outcome assesses the correlation between ultrasound-derived muscle morphology parameters-including muscle thickness, fascicle length, pennation angle, echo intensity, cross-sectional area, stiffness (via shear wave elastography), and vascularity (via microvascular imaging)-and standardized motor function scores (e.g., GMFM-66, GMFCS, MACS, MAS, and Tardieu Scale) in ambulatory children with spastic cerebral palsy.
Comparison Between Modified Heckmatt Scale and Quantitative Echo Intensity in Spastic Muscles | At baseline (single assessment session)
  This outcome evaluates the agreement between visual muscle echogenicity scores based on the Modified Heckmatt Scale and quantitative grayscale echo intensity values obtained via B-mode ultrasonography in spastic upper and lower limb muscles of children with spastic cerebral palsy. The analysis aims to determine the clinical utility of the Modified Heckmatt Scale in representing objective muscle echotexture.

SECONDARY OUTCOMES:
Development of a Composite Muscle Quality Index Based on Ultrasonographic Parameters | At baseline (single assessment session)
  This outcome explores the development of a composite muscle quality scoring system that integrates multiple ultrasonographic parameters-including muscle echo intensity, stiffness (via shear wave elastography), vascularity (via superb microvascular imaging), and architectural features (e.g., muscle thickness, pennation angle, and fascicle length). The aim is to identify a reliable, non-invasive ultrasonographic muscle quality index for characterizing spastic muscles in children with cerebral palsy, potentially guiding future clinical assessment and rehabilitation planning.

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University Faculty of Medicine, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The plan to share individual participant data (IPD) is currently undecided. The study involves pediatric participants with spastic cerebral palsy, and IPD sharing will depend on institutional policies, ethical committee approval, and the extent to which anonymization and parental consent can ensure participant privacy.

REFERENCES:
- [Result] Atalay KG, Saygi EK, Akbas F, Coskun OK, Akgulle AH, Yagci I. Does ultrasound imaging of the spastic muscle have an additive effect on clinical examination tools in patients with cerebral palsy?: A pilot study. North Clin Istanb. 2022 Mar 11;9(2):102-108. doi: 10.14744/10.14744/nci.2020.78045. eCollection 2022. PMID 35582513
- [Result] Peeters N, Hanssen B, Bar-On L, De Groote F, De Beukelaer N, Coremans M, Van den Broeck C, Dan B, Van Campenhout A, Desloovere K. Associations between muscle morphology and spasticity in children with spastic cerebral palsy. Eur J Paediatr Neurol. 2023 May;44:1-8. doi: 10.1016/j.ejpn.2023.01.007. Epub 2023 Jan 10. PMID 36706682
- [Result] Uzun Akkaya K, Akkaya HE, Bezgin S, Atalan Efkere P, Firat T, Yildiz C, Elbasan B. Long-Term Effects of Different Number of Botulinum Toxin Injections Into the Gastrocnemius Muscle on Function and Muscle Morphology in Children With Cerebral Palsy. Pediatr Neurol. 2025 Jan;162:97-104. doi: 10.1016/j.pediatrneurol.2024.10.013. Epub 2024 Oct 22. PMID 39579461
- [Result] Kawano A, Yanagizono T, Kadouchi I, Umezaki T, Chosa E. Ultrasonographic evaluation of changes in the muscle architecture of the gastrocnemius with botulinum toxin treatment for lower extremity spasticity in children with cerebral palsy. J Orthop Sci. 2018 Mar;23(2):389-393. doi: 10.1016/j.jos.2017.10.012. Epub 2017 Nov 14. PMID 29146092
- [Result] Gitto S, Messina C, Chianca V, Tuscano B, Lazzara A, Corazza A, Pedone L, Albano D, Sconfienza LM. Superb microvascular imaging (SMI) in the evaluation of musculoskeletal disorders: a systematic review. Radiol Med. 2020 May;125(5):481-490. doi: 10.1007/s11547-020-01141-x. Epub 2020 Feb 4. PMID 32020529
- [Result] Rosenbaum P, Paneth N, Leviton A, Goldstein M, Bax M, Damiano D, Dan B, Jacobsson B. A report: the definition and classification of cerebral palsy April 2006. Dev Med Child Neurol Suppl. 2007 Feb;109:8-14. PMID 17370477
- See also: Ultrasonographic evaluation of changes in the muscle architecture of the gastrocnemius with botulinum toxin treatment for lower extremity spasticity in children with cerebral palsy — https://pubmed.ncbi.nlm.nih.gov/29146092/